CLINICAL TRIAL: NCT00832728
Title: Safety and Efficacy of the Extracorporeal Liver Assist Device (ELAD®) In Patients With Fulminant Hepatic Failure (FHF)
Acronym: ELAD
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: To focus on another clinical indication.
Sponsor: Vital Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VTI-202
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Fulminant Hepatic Failure
MeSH Terms: conditions — Liver Failure, Acute | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ELAD (Active Comparator): ELAD Therapy + Standard of Care
  Interventions: Other: Standard of Care; Device: ELAD®
- Standard of Care (Other): Hospital based standard of care for acute liver failure
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Standard of Care — Standard hospital protocol for the treatment of acute liver failure
Device: ELAD® — ELAD therapy
  Arms: ELAD

SUMMARY:
This is a multicenter, open-label, randomized, concurrent control study of subjects with FHF. Subjects meeting the eligibility requirements of the study will be randomly assigned in a 2:1 ratio to receive either standard medical therapy for FHF plus the ELAD® system, or standard medical therapy alone, with the latter defined as conventional therapy for FHF determined to be clinically appropriate by the treating physician.

DETAILED DESCRIPTION:
Therapy will generally include treatment of hepatic encephalopathy using lactulose with or without oral antibiotics, antibiotics as indicated to treat infection, volume resuscitation and vasopressors as indicated to treat hypotension. In addition general medical treatment such as glucose control and renal replacement therapy will be used as necessary. Subjects with a clinical diagnosis of hepato-renal syndrome may be treated with midodrine and octreotide or terlipressin, if considered appropriate therapy.

Immediately prior to treatment initiation, subject eligibility will be confirmed. Treatment with ELAD® will continue for a minimum of 3 days and up to a maximum of 30 days, until, in the Investigator's opinion, clinical status improves relative to entry; until the subject undergoes OLT; or until the continued use of ELAD® is contraindicated, as described in Section 5.5. Subjects will be followed until discontinuation or 30 days has elapsed since study enrollment (control) or 30 days has elapsed since cessation of ELAD® therapy (ELAD® group), whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Weight ≥15 kilograms;
2. Age ≥10 ≤65 years;
3. Diagnosis of FHF;
4. Patients must have been treated with a standard regimen of N-acetyl cysteine (NAC) involving a loading dose of 150mg/kg/hr over 1 hour followed by 12.5 mg/kg/hour x 4 hours then continuous infusion of 6.25 mg/kg for the remaining 67 hrs.
5. Subject or designated representative must be willing to sign an Informed Consent Form specific to this study and comply with study requirements AND EITHER
6. Known acetaminophen ingestion or diagnostic serum level, and at least one of the following:

   a. prothrombin time (PT) >30 seconds (International Normalized Ratio (INR) >6.5, OR; b. Encephalopathy Grade II, III or IV and at least one of the following: i. Arterial pH <7.30 at ≥2 hours after initial diagnosis, OR; ii. renal failure documented by urine output less than 2 mL/kg/hr over 12 hours, OR; iii. creatinine >2.5 mg/dL; OR
7. Patients with Non-Acetaminophen-Induced FHF:

   a. Stage II, III or IV encephalopathy, and the presence of at least two of the following five criteria: i. Non-A/Non-B hepatitis or drug (non-acetaminophen) induced FHF; ii. Serum bilirubin >17 mg/dL; iii. Patient ≥10 or <40 years old; iv. Prothrombin time >25 seconds (INR > 3.5), AND/OR; v. Jaundice to encephalopathy time ≥7 days; OR
8. Liver transplantation within 10 days of the screening procedures, but meeting inclusion criteria due to primary graft non-function, and not receiving ELAD® therapy prior to the first graft

Exclusion Criteria:

1. Cerebral Perfusion Pressure as measured by an intracranial pressure (ICP) monitor. (NOTE: In those cases where ICP monitor placement cannot be performed prior to study enrollment, this exclusion criterion will not apply):

   1. Patients > 18 yrs of age with Cerebral Perfusion Pressures (CPP) ≤40 mm Hg for one hour or longer.
   2. Patients ≤18 yrs with CPP ≤35 mm Hg for one hour or longer.
2. Chronic liver disease;
3. Concomitant disease including chronic congestive heart failure, vascular disease, emphysema, AIDS, cancer, acute fatty-liver disease, hepatitis due to herpes virus, Wilson's disease, or Budd-Chiari syndrome;
4. Portal hypertension (e.g., variceal bleed, caput Medusae, and clinically obvious ascites);
5. Liver dysfunction due to trauma;
6. Hemorrhage or irreversible brain death ( i.e. blood flow studies positive for herniation and/or pupillary reflex absent);
7. Platelet count <50,000/mm3 or reducing to <80,000/mm3 over a 72 hr. period. (NOTE: Patient may be included at the physician's discretion if platelet count exceeds 50,000mm3 at time of initiation of therapy and can be managed through the administration of blood products);
8. Mean Arterial Pressures (MAP) ≤50 mm Hg for one hour or longer as measured by an indwelling arterial line, OR; patients ≤18 years old and whose MAP is ≤40 mm Hg for one hour or longer;
9. Vasopressor support exceeding 1.0 µg/kg/min of an alpha-adrenergic agent for one hour or longer;
10. Clinical or radiographic evidence of stroke or intracerebral bleeding;
11. Seizures uncontrolled by medication;
12. Acute myocardial infarction based on clinical and/or electrocardiographic evidence;
13. Lung disease defined by a PaO2 ≤ 60mm Hg or an FiO2 ≥0.6, not corrected by medical management (including CVVH if indicated);
14. Pregnancy as determined by βhCG results;
15. ≤2 weeks postpartum;
16. Participation in another investigational study within 30 days of enrollment;
17. Prior ELAD® therapy.

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The effect of ELAD® therapy: 1) as a bridge-to-transplant/recovery and 2) on 30-day transplant-free survival in subjects with FHF | 30 day
To assess its safety when used for a minimum of 3 days or up to a maximum of 30 days of treatment | 30 day

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Ashley, Study Director — Vital Therapies, Inc.
Locations (12):
- United States (12):
  - Scripps Green Hospital, La Jolla, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - Loyola University Medical Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Louisiana State University Health Sciences Center-Shreveport, Shreveport, Louisiana
  - New York University Medical Center, New York, New York
  - University of Rochester, Strong Memorial, Rochester, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia